CLINICAL TRIAL: NCT06491225
Title: A Phase I, Open Label, Multicenter Study Evaluating the Safety and Efficacy of Autologous Tumor-Infiltrating Lymphocyte (GTE-001 Injection ) for Treatment of Patients with Advanced Lung Adenocarcinoma
Brief Title: Autologous Tumor-Infiltrating Lymphocyte (GTE-001 Injection ) for Treatment of Patients with Advanced Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTE-001-001
Record Dates: First submitted 2024-06-30; First posted 2024-07-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Advanced Lung Adenocarcinoma；Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GTE001 injection treatment group (Experimental)
  Interventions: Biological: GTE001 injection

INTERVENTIONS:
Biological: GTE001 injection — GTE-001 injection to treat Advanced lung adenocarcinoma

SUMMARY:
This study is a Multiple centers, open design aimed at evaluating the safety,efficacy and Production feasibility of Autologous Tumor-Infiltrating Lymphocyte (GTE-001 injection ) for treatment of patients with Advanced lung adenocarcinoma,And evaluate potential biomarkers related to GTE-001 activity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily join the study, signed informed consent form， willing and able to comply with the study protocol;
* 2. Age ≥18 years old;
* 3. Advanced lung adenocarcinoma that progresses after recurrence or first-line chemotherapy；
* 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* 5. Expected survival time of ≥ 3 months;
* 6. Good function of vital organs;
* 7. At least one measurable target lesion that meets the definition of RECIST v1.1 after tumor sampling.

Exclusion Criteria:

* 1.Subject has previously received an allogeneic stem cell transplant or organ allograft,Subject has previously received engineered cell therapy,Prior FOLR1 directed therapy is not allowed unless it had been with an approved agent in the indication;
* 2.Subject has undergone surgery or received radiotherapy, immunotherapy, targeted therapy agents, anticancer vaccines, systemic steroids, or chemotherapy within 2 weeks of enrolment. Targeted agents, such as tyrosine kinase inhibitors, may be continued until 5 half-lives before enrolment;
* 3.Pregnant or lactating women; or women who are pregnant, breastfeeding, or planning to become pregnant within 12 months after cell infusion;
* 4.History of central nervous system (CNS) disorder,History of autoimmune disease,History of primary immunodeficiency;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-07-18 (Estimated); Study Completion 2027-07-18 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 years
  To evaluate efficacy parameters such Objective Response Rate (ORR) per RECIST 1.1, as assessed by the Investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No